CLINICAL TRIAL: NCT06226857
Title: Predictive Value of Other Oncogene Mutations for Anti-EGFR Monoclonal Antibodies Efficacy in Patients With Left-sided RAS-wild Type Metastatic Colorectal Cancer: Multicenter Randomized Phase III Trial
Brief Title: Other Oncogene Mutations for Anti-EGFR Efficacy in Patients With Left-sided RAS-wild Type Metastatic Colorectal Cancer
Acronym: CRC01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: City Clinical Oncology Hospital No 1 (Other Government)
Collaborators: Atlas Biomed (Industry); N.N. Blokhin National Medical Research Center of Oncology (Other); Moscow MultidisciplinaryClinical Center Kommunarka (Unknown)
Responsible Party: Principal Investigator, Pokataev Ilya, Head of department of medical oncology, City Clinical Oncology Hospital No 1
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRC01; 2102-2/23 (Other Grant/Funding Number: Moscow Center for healthcare innovations)
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Neoplasms; Chemotherapy Effect; Molecular Sequence Variation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Panitumumab

STUDY DESIGN:
Intervention Model Description: randomize and compare contol and experimental groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Active Comparator): All patients will recieve chemotherapy FOLFOX (oxaliplatin 85 mg/m2 + folinic acid 400 mg/m2 + FU 400 mg/m2 bolus and FU 2400 mg/m2 46-hour insusion q2w) + anti-EGFR monoclonal antibody (cetuximab 500 mg/m2 q2w or panitumumab 6 mg/kg q2w) until disease progression or unacceptable toxicity. It is permited to withdraw oxaliplatin after 8 cycles.
  Interventions: Drug: Cetuximab
- BC (Experimental): All patients will recieve chemotherapy FOLFOX (oxaliplatin 85 mg/m2 + folinic acid 400 mg/m2 + FU 400 mg/m2 bolus and FU 2400mg/m2 46-hour insusion q2w). Monoclonal antibody will be added to chemotherapy after 1-2 cycles based on molecular profile results: anti-EGFR (cetuximab 500 mg/m2 q2w or panitumumab 6 mg/kg q2w) for hyperselected wild type tumors or bevacizumab 5 mg/m2 q2w for mutant profile.
  Patients will recieve therapy until disease progression or unacceptable toxicity. It is permited to withdraw oxaliplatin after 8 cycles.
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — FOLFOX+cetuximab/panitumumab q2w until desease progression, deescalation to de Gramont+cetuximab/panitumumab is allowed after 8 cycles
  Other Names: panitumumab

SUMMARY:
Patients meeting the inclusion criteria will be randomized 1:1 into Cohort A (n ≈ 177) or Cohort BC (n ≈ 177). Cohort A is the control: patients receive combination chemotherapy with FOLFOX plus anti-EGFR therapy (panitumumab or cetuximab) based on RAS/BRAF wild-type data, according to clinical guidelines.

The BC cohort begins FOLFOX chemotherapy and simultaneously undergoes extensive molecular genetic profiling. Further, the BC cohort, depending on the profile, is divided into cohort B - patients without changes in alternative oncogenes, and cohort C - with changes in alternative oncogenes. The expected cohort ratio is 3:1 (~120 and ~40 patients). Cohort B begins to receive anti-EGFR therapy in addition to chemotherapy, and the potentially resistant cohort C continues to receive chemotherapy alone or begins to receive bevacizumab if there are no contraindications.

DETAILED DESCRIPTION:
In total, the study plans to include 355 patients diagnosed with unresectable metastatic colorectal cancer with a left-sided localization of the primary tumor, who have not previously received systemic therapy for metastatic disease, have wild-type KRAS/NRAS/BRAF, or have wild-type KRAS/NRAS with unknown BRAF status in no contraindications to targeted therapy (cetuximab/panitumumab/bevacizumab).

Patients meeting the inclusion criteria will be randomized 1:1 into Cohort A (n ≈ 177) or Cohort BC (n ≈ 177). Cohort A is the control: patients receive combination chemotherapy with FOLFOX plus anti-EGFR therapy (panitumumab or cetuximab) based on RAS/BRAF wild-type data, according to clinical guidelines. Next, this cohort, after completion of the protocol, undergoes extended profiling, according to the results of which it is divided into cohorts A1 and A2. Cohort A1 includes patients without changes in alternative oncogenes (N ≈ 120), cohort A2 includes patients with changes (N ≈ 40).

The BC cohort begins FOLFOX chemotherapy and simultaneously undergoes extensive molecular genetic profiling. Further, the BC cohort, depending on the profile, is divided into cohort B - patients without changes in alternative oncogenes, and cohort C - with changes in alternative oncogenes. The expected cohort ratio is 3:1 (~120 and ~40 patients). Cohort B begins to receive anti-EGFR therapy in addition to chemotherapy, and the potentially resistant cohort C continues to receive chemotherapy alone or begins to receive bevacizumab if there are no contraindications.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed before commencing any procedures related to the clinical trial.
2. Age ≥18 years.
3. ECOG status 0-2.
4. Life expectancy greater than 12 weeks as assessed by the investigator.
5. Verified diagnosis of colorectal adenocarcinoma (C18.5, C19, C20).
6. Metastatic unresectable form of the disease that has not previously received any systemic therapy for the metastatic process (previous neo-/adjuvant therapy completed at least 6 months before the detection of metastases is allowed).
7. Left-sided localization of the primary tumor (from the splenic flexure of the colon inclusive).
8. Verified wild type KRAS, NRAS determined from tumor tissue.
9. Satisfactory function of hematopoiesis and internal organs:

   * absolute number of neutrophils ≥ 1.5×10 9 /l;
   * platelets ≥ 100×10 9 /l;
   * hemoglobin ≥ 90 g/l.
   * creatinine clearance above 50 ml/min;
   * total bilirubin <1.5 X the upper limit of normal;
   * ALT or AST >5 X the upper limit of normal in the presence of liver metastases or >2.5 X the upper limit of normal in the absence of liver metastases.
10. Availability of a sufficient amount of tumor material for molecular genetic research. Tumor material must be collected no more than 24 months before inclusion in the study.

Exclusion Criteria:

1. Previous systemic therapy for metastatic disease.
2. Presence of KRAS/NRAS/V600E mutations (except for unknown BRAF status).
3. Uncertain KRAS/NRAS status
4. The presence of any other malignant tumor, with the exception of radically treated basal cell carcinoma, cervical cancer in situ, currently or within 5 years before inclusion in the study. Pregnant and lactating women, as well as planning pregnancy during the period of therapy in a clinical trial and 6 months after the end of therapy.
5. HIV infection, active hepatitis B, active hepatitis C.
6. Complicated primary tumor, requiring urgent surgical intervention. After it is eliminated, the patient can participate in the study.
7. The presence of a disease or condition that, in the opinion of the investigator, prevents the patient from participating in the study.
8. Impossibility of organizing central venous access.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | through study completion, an average of 3 years
  Intention to treat, Calculated from start of therapy to date of disease progression or death

SECONDARY OUTCOMES:
edverse events | through study completion, an average of 3 years
  all AE based on CTC criteria v. 5
overall survival | through study completion, an average of 3 years
  Calculated from start of therapy to date of last contact or death
progression-free survival based (per protocol) | through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Moscow Multidiciplinary Clinical Center Kommunarka, Moscow
  - N.N Blokhin Cancer Reserch Center, Moscow
  - Reutov Clinical hospital, Reutov

IPD SHARING:
Plan to Share IPD: Undecided